CLINICAL TRIAL: NCT05030714
Title: Evaluation of a Novel Head-Mounted Device for Glaucoma Testing: A Proof-of-Concept Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brennan Eadie (Other)
Responsible Party: Sponsor-Investigator, Brennan Eadie, Assistant Professor, Department of Ophthalmology, Dalhousie University and Nova Scotia Health Authority; MD, PhD, FRCSC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E002
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Visual Fields

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will perform visual field testing with the Humphrey Visual Field Analyzer and with the custom head-mounted device.
  Interventions: Diagnostic Test: Visual Field Testing

INTERVENTIONS:
Diagnostic Test: Visual Field Testing — Visual field testing using the protocol 24-2 and/or 10-2 Threshold Test

SUMMARY:
This proof-of-concept study aims to determine the feasibility and effectiveness of using a custom head-mounted device for visual field testing. The novel head-mounted device, with custom software, will be compared to a conventional visual field test: The Humphrey Visual Field Analyzer. The investigators will include 30 healthy normal patients, 30 glaucoma suspects, 30 patients with moderate glaucoma, and 30 patients with advanced glaucoma (total: 120 patients). Each patient will perform the conventional test and the head-mounted device visual field test during the study visit, with the order (i.e., which device the patient starts with) being randomized. After the two tests, the patient will fill out a questionnaire to gather information regarding patient comfort and satisfaction. This will repeat each week for 5 weeks, for a total of 5 study visits. The results of the tests (sensitivity thresholds) will be compared. The investigators hypothesize that the results of the conventional and head-mounted device will be similar.

ELIGIBILITY:
Inclusion Criteria:

* Previous visual field test with Humphrey Field Analyzer indicating normal field, early glaucomatous field damage, moderate glaucomatous field damage, or advanced glaucomatous field damage.
* Ability to understand and consent to the study.

Exclusion Criteria:

* Diagnosis of secondary glaucoma
* Diagnosis of non-glaucomatous optic neuropathy or other significant ophthalmic diagnosis that could limit vision (ex. age-related macular degeneration)
* Significant media opacity
* Previous intraocular surgery other than cataract surgery
* Anxiety disorder
* Pregnancy
* Seizure disorder
* Cardiac pacemaker or other implantable devices
* Severe vertigo or balance disturbance
* Refractive error greater than +4 diopters and less than -6 diopters spherical equivalent
* Inability to demonstrate competence to make informed decision regarding study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Visual field differential light sensitivity | 5 weeks
  Comparison of differential light sensitivity threshold estimated with the Humphrey Visual Field Analyzer and the custom head-mounted device.

SECONDARY OUTCOMES:
Reproducibility of sensitivity values | 5 weeks
  Comparison of the reproducibility of sensitivity values estimated with the Humphrey Visual Field Analyzer and the custom head-mounted device.

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Eadie, MD, PhD, Principal Investigator — Nova Scotia Healthy Authority
Locations (2):
- Canada (2):
  - Victoria General Hopsital - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Eadie Technologies Inc., Halifax, Nova Scotia